CLINICAL TRIAL: NCT05284279
Title: Early Childhood Caries and Health Professionals' Perception: a Qualitative Research Protocol to Assess Oral Health Stigma
Acronym: CariStigma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_1182
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Early Childhood Caries (ECC)
Keywords: Dental caries; Social stigma; child; qualitative study
MeSH Terms: conditions — Dental Caries; Social Stigma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health professionals practicing with children: To participate, health professionals will have to speak French fluently, practice with children as a dentist (general or pediatric), a general practitioner, or a paediatrician and work in hospital or ambulatory facility. As paediatricians and general practitioners meet the child regularly during the first 6 years of life for medical follow-up, they are key stakeholders in the early detection of caries, referrals to dentist and counselling.
  The participants will be recruited using a semi-random sampling method. The sample will be constituted with a maximum variation in age, gender, years in practice, occupation and types of practice (solo, group or interdisciplinary team).
  Interventions: Other: Exploring health professionals' perceptions of patients with ECC using semi-structured interviews

INTERVENTIONS:
Other: Exploring health professionals' perceptions of patients with ECC using semi-structured interviews — Following a literature review on the topic of children with ECC and their family, a guidebook will be built by main investigators. Several test interviews will be conduct to ensure that guidebook is adapted, and that the interviewer is enough trained.
  Interview will be conducted by one or two of the main investigators. As much as possible, they will be performed face to face or using videoconference due to COVID19 pandemic context. All the interviews will be audio recorded. The interviewer will take notes including non-verbal communication; and will adopt an active listening position.
  After collecting respondents' characteristics (age, gender, profession, exercise duration, type of practice), the subsequent themes will be explored: disease perception, educational context's responsibility, barriers and facilitators to family behaviour changes, health professional's emotional consequences.

SUMMARY:
Dental caries is the most common non-communicable disease in childhood. Disease management of caries rests on surgical treatment as well as various preventive strategies such as fluoridation, sealants, personal counselling...

With other non-communicable diseases (obesity, overweight…), it has been demonstrated that health professionals' negative perceptions of their patients could affect disease management quality. Concerning dental caries, some data might suggest that discriminating believes and behaviours toward children with dental caries and their families exist in the medical setting. However, oral health related stigma remains an unexplored issue. This study would be the first to our knowledge to specifically address the question of stigmatisation and discrimination of patients with dental caries. The present project is to conduct an exploratory study focusing on perceptions and attitudes of health professionals toward children with early childhood caries and their parents.

The questions the study aims to answer are: (i) What are health professionals 'perceptions of children with ECC and their family? And (ii) according to health professionals, do these perceptions influence the quality of their care? We hypothesize that some practitioners have negative opinions on children with ECC and their parents, affecting the quality of their care, especially concerning oral health prevention.

Method: Individual semi-structured interviews will be conducted among dentists (general or pediatric), general practitioners and paediatricians.

ELIGIBILITY:
Inclusion Criteria:

* speak French fluently
* practice with children as a dentist (general or pediatric), a general practitioner, or a paediatrician
* work in hospital or ambulatory facility

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants' selection will be conducted on a semirandom basis, directly from the network of the research team members and from regional professional listings of each specialty (general practitioners, pediatricians, general dentists, pediatric dentists). The sample will be constituted with a maximum variation in age, gender, years in practice, occupation and types of practice (solo, group or interdisciplinary team).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Health professionals' representations of children with dental caries and their family | The main outcome will be collected during the interviews.
  Individual semi-structured interviews will be conducted among dentists, general practitioners and paediatricians to explore health professionals' representations of children with dental caries and their family. All the interviews will be audio recorded and transcribed into verbatims. Verbatims will be analysed using the N'Vivo qualitative analysis software. The thematic analysis of the data will then be carried out using the 6-steps method of Braun and Clarke. A transversal analysis will be conducted by classifying the verbatims of each interview into themes and main theme.

CONTACTS AND LOCATIONS:
Locations (1):
- As much as possible, interviews will be performed face to face at a location convenient to the respondent or using videoconference due to COVID19 pandemic context., Rhone-Alpes Region, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lienhart G, Thivichon-Prince B, Farge P, Schott-Pethelaz AM, Chaneliere M. What are health professionals' perceptions and attitudes regarding children with early childhood caries and their families? A qualitative research protocol to assess oral health stigma in the medical setting. BMJ Open. 2022 Dec 1;12(12):e066680. doi: 10.1136/bmjopen-2022-066680. PMID 36455999